CLINICAL TRIAL: NCT00044018
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Two CDC-501 Dose Regimens When Used Alone or in Combination With Dexamethasone for the Treatment Relapsed or Refractory Multiple Myeloma
Brief Title: CDC-501 Therapy in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-007
Record Dates: First submitted 2002-08-16; First posted 2002-08-20 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Revimid; CC5013
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CDC-501

SUMMARY:
The purpose of the study is to select the dose regimen of CDC-501 that provides the most promising evidence of efficacy.

ELIGIBILITY:
* Subject must be diagnosed with multiple myeloma (with measurable M-Protein in serum and/or urine), and be considered to have disease progression after at least two cycles of treatment or have relapsed after treatment.
* Subject must understand and voluntarily sign an informed consent document.
* Subject must not have received corticosteroids, other chemotherapy, thalidomide, or other investigational agents, within 21 days of baseline
* ECOG (Zubrod) performance status of 0 to 2.
* Subject must be able to adhere to the study visit schedule and other protocol requirements.
* Women of childbearing potential (WCBP ) must have a negative serum or urine pregnancy test within 7 days of baseline. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2002-04-01 (Actual); Primary Completion 2004-12-01 (Actual); Study Completion 2007-02-15 (Actual)

PRIMARY OUTCOMES:
Confirmed M-Protein Response During Single Agent CDC-501 Therapy | Response assessed every 4 weeks; up to 62 months
  M-Protein response evaluated every 4 weeks through urine and serum electrophoresis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (4):
- United States (4):
  - H Lee Moffit Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - St Vincent's Cancer Center, New York, New York

REFERENCES:
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727